CLINICAL TRIAL: NCT05840523
Title: The Effect of Hip Abductor Strengthening With Proprioceptive Neuromuscular Facilitation and Elastic Resistive Band Exercises on Core Endurance and Functional Performance ın Healthy Adults
Brief Title: Hip Abductor Strengthening With Proprioceptive Neuromuscular Facilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Feyza Altındal, Assistant Professor, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NigdeFAltındal
Record Dates: First submitted 2022-08-31; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Sports Physical Therapy
Keywords: Exercise; Muscle strenght; Balance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into three groups using the sealed envelope method (on the evaluation day, participants chose one of the sealed envelopes and determined the treatment group). Group I comprised the Proprioceptive Neuromuscular Facilitation (PNF) group, Group II the Range of Motion(ROM) group, and Group III the Control (CG) group. Evaluations were made at baseline and at sixth week.
Who Masked: Participant
Masking Description: Participants were randomly divided into three groups using the sealed envelope method (on the evaluation day, participants chose one of the sealed envelopes and determined the treatment group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Neuromuscular Facilitation (PNF) Exercise Group (Experimental): The PNF group performed flexion-abduction-internal rotation and extension-abduction-internal rotation patterns as 15 repetitions, 2 sets. The metronome was used to fix the construction speed of the exercises (50bpm). PNF exercises were performed with EB at a metronome speed of 50bpm at a ratio of 1:2 sec. In other words, while transition from the antagonist to agonist pattern in 3 clicks, there was return from agonist to antagonist in 6 clicks.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation exercises
- Range Of Motion (ROM) Exercise Group (Experimental): The ROM group performed hip flexion abduction, neutral abduction and extension abduction exercises with an EB at 50bpm metronome speed in 3 sets of 10 repetitions. In both groups, 30 seconds of rest was given between exercises.
  Interventions: Other: The Range Of Motion exercises
- Control Group (No Intervention): No exercise practice was done

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation exercises — The PNF group performed flexion-abduction-internal rotation and extension-abduction-internal rotation patterns as 15 repetitions, 2 sets. The metronome was used to fix the construction speed of the exercises (50bpm). PNF exercises were performed with EB at a metronome speed of 50bpm at a ratio of 1:2 sec. In other words, while transition from the antagonist to agonist pattern in 3 clicks, there was return from agonist to antagonist in 6 clicks.
  Arms: Proprioceptive Neuromuscular Facilitation (PNF) Exercise Group
Other: The Range Of Motion exercises — The ROM group performed hip flexion abduction, neutral abduction and extension abduction exercises with an EB at 50bpm metronome speed in 3 sets of 10 repetitions. In both groups, 30 seconds of rest was given between exercises.
  Arms: Range Of Motion (ROM) Exercise Group

SUMMARY:
Objectives: To compare effectiveness of strengthening hip abductors with Proprioceptive Neuromuscular Facilitation (PNF) technique and Range Of Motion (ROM) exercises on core endurance and functional performance in healthy adults using theraband.

Methods: 66 sedentary healthy, male volunteers between ages 20-26 (mean age 21,68± 1,37 years) participated in study. PNF, ROM exercises applied with theraband include intervention groups. Theraband strengthening exercises were applied 3 days a week for 6 weeks, a total of 18 sessions. Intervention groups were compared with healthy control group. Participants hip abductor muscle strength was assessed with hand held dynamometer, lower extremity balance with y test, core endurance with flexor, extensor, right, left side endurance tests, global core stability with single leg squat test at baseline and at 6 weeks after exercise program.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial and conducted according to the Declaration of Helsinki and was approved by the Ethics Committee of Clinical Trials (21.05.2019/10). All participants were informed about the study and their written consent was obtained. Participants were randomly divided into three groups using the sealed envelope method (on the evaluation day, participants chose one of the sealed envelopes and determined the treatment group). Group I comprised the Proprioceptive Neuromuscular Facilitation (PNF) group, Group II the Range of Motion(ROM) group, and Group III the Control (CG) group. Evaluations were made at baseline and at sixth week. Male participants between the ages of 20 and 26 years, were included in the study. Participants age, body mass index (BMI), dominant extremity were recorded as descriptive data.

Muscle strength assessment: Bilateral hip abductor isometric strength was assessed using a Hand-held Dynamometer (HHD) (Commander Power Track II; JTECH Medical Industries, Salt Lake City, UT) using the maximal isometric strength standard protocol. The participant was asked to 30 degree hip abduct by stabilizing the pelvis in the side lying position. Three measurements were made by placing the dynamometer pad 10 cm proximal to the lateral epicondyle of the femur, and the average value was recorded in kilograms.

Balance assesment: It was done with Y balance test. While maintaining their balance on the dominant extremity on the test platform, the participants were asked to reach out in 3 directions (anterior-posterior, postero-medial and postero-lateral) with the tip of the other foot. 3 repetitions were made for each direction, and rest intervals of 15 seconds were given. The mean score was recorded in cm. The lower extremity length of the participants was determined by measuring the distance between the anterior superior spina iliaca and the medial malleolus with a tape measure in the supine position. Composite scoring was obtained by multiply with one hundred the reach in all directions and dividing by three leg lengths.

Global (functional) core assessment: It was done with the single leg squat test. Participants were asked to perform one-leg squats at 45 degree knee flexion in 30 seconds, and the number of squats was recorded.

Core endurance assessment: Participants were evaluated with trunk flexion endurance, extension endurance and lateral bridge endurance tests, and the results were recorded in seconds.

ELIGIBILITY:
inclusion criteria:

* Not having any known and diagnosed health problems
* Not exercising regularly
* Not having a lower/upper extremity injury in the last three months
* Volunteering to participate in the study

exclusion criteria:

* Not to participate in exercise training more than three sessions
* Want to leave the training voluntarily
* Have experienced serious orthopedic/systemic discomfort during the training

Ages: 20 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Muscle strength with different exercises(PNF and ROM) at week 6 | 6 weeks
  Bilateral hip abductor isometric strength was assessed using a Hand-held Dynamometer(HHD) (Commander Power Track II; JTECH Medical Industries, Salt Lake City, UT) using the maximal isometric strength standard protocol. The participant was asked to 30 degrees hip abduct by stabilizing the pelvis in the side lying position. Three measurements were made by placing the dynamometer pad 10 cm proximal to the lateral epicondyle of the femur, and the average value was recorded in kilograms.
Change from baseline in balance with different exercises(PNF and ROM) at week 6 | 6 weeks
  It was done with Y balance test. While maintaining their balance on the dominant extremity on the test platform, the participants were asked to reach out in 3 directions (anterior-posterior, postero-medial and postero-lateral) with the tip of the other foot. 3 repetitions were made for each direction, and rest intervals of 15 seconds were given. The mean score was recorded in cm. The lower extremity length of the participants was determined by measuring the distance between the anterior superior spina iliaca and the medial malleolus with a tape measure in the supine position. Composite scoring was obtained by multiply with one hundred the reach in all directions and dividing by three leg lengths.
Change from baseline in global(functional) core with different exercises(PNF and ROM) at week 6 | 6 weeks
  It was done with the single leg squat test. Participants were asked to perform one-leg squats at 45 degrees knee flexion in 30 seconds, and the number of squats was recorded.
Change from baseline in core endurance with different exercises(PNF and ROM) at week 6 | 6 weeks
  Participants were evaluated with trunk flexion endurance, extension endurance and lateral bridge endurance tests, and the results were recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Büker, Prof. Dr, Study Director — Pamukkale Üniversity Physical Theraphy and Rehabilitation Faculty TURKEY; Feyza Altındal, PhD, Principal Investigator — Niğde Ömer Halisdemir Üniversity Physical Theraphy and Rehabilitation Departmant TURKEY
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SP, Powers CM. Individuals with diminished hip abductor muscle strength exhibit altered ankle biomechanics and neuromuscular activation during unipedal balance tasks. Gait Posture. 2014 Mar;39(3):933-8. doi: 10.1016/j.gaitpost.2013.12.004. Epub 2013 Dec 12. PMID 24373699
- [Background] Park KM, Kim SY, Oh DW. Effects of the pelvic compression belt on gluteus medius, quadratus lumborum, and lumbar multifidus activities during side-lying hip abduction. J Electromyogr Kinesiol. 2010 Dec;20(6):1141-5. doi: 10.1016/j.jelekin.2010.05.009. Epub 2010 Jun 19. PMID 20646935
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] Boling M, Padua D. Relationship between hip strength and trunk, hip, and knee kinematics during a jump-landing task in individuals with patellofemoral pain. Int J Sports Phys Ther. 2013 Oct;8(5):661-9. PMID 24175145
- [Background] Song HS, Park SD, Kim JY. The effects of proprioceptive neuromuscular facilitation integration pattern exercise program on the fall efficacy and gait ability of the elders with experienced fall. J Exerc Rehabil. 2014 Aug 31;10(4):236-40. doi: 10.12965/jer.140141. eCollection 2014 Aug. PMID 25210699
- [Background] Pozzi F, White DK, Snyder-Mackler L, Zeni JA. Restoring physical function after knee replacement: a cross sectional comparison of progressive strengthening vs standard physical therapy. Physiother Theory Pract. 2020 Jan;36(1):122-133. doi: 10.1080/09593985.2018.1479475. Epub 2018 Jun 7. PMID 29877749
- [Background] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Rhyu HS, Kim SH, Park HS. The effects of band exercise using proprioceptive neuromuscular facilitation on muscular strength in lower extremity. J Exerc Rehabil. 2015 Feb 28;11(1):36-40. doi: 10.12965/jer.150189. eCollection 2015 Feb. PMID 25830142
- [Background] 17. Kang DH, Lee WH, Lim S, Kim YY, An SW, Kwon CG, Lee GH, Choi NR, Lee NY, Kim BM, Kim JH, Chung EJ. The effect of hip joint exercise using an elastic band on dynamic balance, agility and flexibility in healthy subjects: a randomized controlled trial Phys Ther Rehabil Sci 2016; 5(4):198-204.
- [Background] Gottlieb GL, Agarwal GC. Modulation of postural reflexes by voluntary movement. II. Modulation at an inactive joint. J Neurol Neurosurg Psychiatry. 1973 Aug;36(4):540-6. doi: 10.1136/jnnp.36.4.540. PMID 4354398
- [Background] 20. Adler S, Beckers D, Buck M: PNF in practice, Springer, Berlin, 2008, s.127-162.
- [Background] Jakobsen MD, Sundstrup E, Andersen CH, Aagaard P, Andersen LL. Muscle activity during leg strengthening exercise using free weights and elastic resistance: effects of ballistic vs controlled contractions. Hum Mov Sci. 2013 Feb;32(1):65-78. doi: 10.1016/j.humov.2012.07.002. Epub 2012 Dec 8. PMID 23231756
- [Background] 22. Kofotolis N, Kellis E. Cross-training effects of a proprioceptive neuromuscular facilitation exercise programme on knee musculature. Phys Ther Sport 2007; 8: 109-116.
- [Background] Ju SK, Yoo WG. Comparison of anterior gluteus medius fiber activation during general exercises and PNF exercises. J Phys Ther Sci. 2017 Mar;29(3):476-477. doi: 10.1589/jpts.29.476. Epub 2017 Mar 22. PMID 28356634
- [Background] 24. DiMattia MA, Livengood AL, Uhl TL, Mattacola CG, Malone TR. What Are the Validity of the Single-Leg-Squat Test and Its Relationship to Hip-Abduction Strength? J Sport Rehabil 2005; 14 (2): 108-123.
- [Background] DeFOREST BA, Cantrell GS, Schilling BK. Muscle Activity in Single- vs. Double-Leg Squats. Int J Exerc Sci. 2014 Oct 1;7(4):302-310. doi: 10.70252/MXVZ7653. eCollection 2014. PMID 27182408
- [Background] Wilson BR, Robertson KE, Burnham JM, Yonz MC, Ireland ML, Noehren B. The Relationship Between Hip Strength and the Y Balance Test. J Sport Rehabil. 2018 Sep 1;27(5):445-450. doi: 10.1123/jsr.2016-0187. Epub 2018 Jul 20. PMID 28714790
- [Background] Ambegaonkar JP, Mettinger LM, Caswell SV, Burtt A, Cortes N. Relationships between core endurance, hip strength, and balance in collegiate female athletes. Int J Sports Phys Ther. 2014 Oct;9(5):604-16. PMID 25328823